CLINICAL TRIAL: NCT00564408
Title: Experimental Study That Investigates the Effect of an Acetylcholine Analogue in Terms of Headache and Changes in Intra- and Extra-cerebral Vessels During and After Infusion of Carbachol
Brief Title: Carbachols Headache-inducing Effect and Changes in Cerebral Blood Flow in Migraine Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Henrik Schytz/MD, Danish HC
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HC20070049
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Carbachol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental)
  Interventions: Drug: Carbachol

INTERVENTIONS:
Drug: Carbachol — 3 microgram per kg bodyweight infused intravenously

SUMMARY:
The purpose of this study is to test if carbachol infusion induces headache in migraine subjects as well as intra- and extra-cerebral vasodilatation.

DETAILED DESCRIPTION:
To test if infusion of Carbachol induces headache in 12 migraine subjects as well as intra- and extra-cerebral vasodilatation in a double-blinded study

ELIGIBILITY:
Inclusion Criteria:

* Migraine without aura
* Weight 50-100 kg

Exclusion Criteria:

* Other significant diseases
* Migraine 5 days prior to experiment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-10 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Headache response after Carbachol infusion | 1 day after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Schytz, MD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark